CLINICAL TRIAL: NCT04003623
Title: A Phase 2, Open-Label, Single-Arm, Multicenter Study to Evaluate the Efficacy and Safety of Pemigatinib in Participants With Previously Treated Locally Advanced/Metastatic or Surgically Unresectable Solid Tumors Harboring Activating FGFR Mutations or Translocations (FIGHT-208)
Brief Title: Efficacy and Safety of Pemigatinib in Participants With Solid Tumors With FGFR Mutations or Translocations (FIGHT-208)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The study was closed due to lack of enrollment.
Sponsor: Incyte Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: INCB 54828-MA-TA-208
Record Dates: First submitted 2019-06-25; First posted 2019-07-01 (Actual); Results first posted 2022-04-21 (Actual); Last update posted 2022-05-10 (Actual); Status verified 2022-04

CONDITIONS: Advanced or Metastatic Solid Tumors; FGFR Mutations; FGFR Translocations
Keywords: Advanced solid tumor; metastatic solid tumor; FGFR inhibitor; FGFR mutation; FGFR translocation
MeSH Terms: conditions — Neoplasm Metastasis | interventions — pemigatinib

STUDY DESIGN:
Intervention Model Description: Participants will be assigned to 1 of 2 cohorts (Cohort A: FGFR1-3 in-frame fusions or FGFR2 intron 17 rearrangements; Cohort B: Known/predicted activating point mutations in FGFR1-3 [excluding kinase domain]) but there is no difference in the treatment regimen between the cohorts.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Pemigatinib (Experimental)
  Interventions: Drug: Pemigatinib

INTERVENTIONS:
Drug: Pemigatinib — Pemigatinib administered orally once daily.
  Other Names: INCB054828

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of pemigatinib in participants with previously treated locally advanced/metastatic or surgically unresectable solid tumors harboring activating FGFR mutations or translocations.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed solid tumor malignancy that is advanced or metastatic (Stage IIIB or IV) or is surgically unresectable.
* Radiographically measurable disease (per RECIST v1.1 or RANO for primary brain tumors).
* Documentation of an FGFR1-3 gene mutation or translocation.
* Objective disease progression after at least 1 prior therapy.
* Not eligible or able to participate in any other Incyte-sponsored clinical trial.

Exclusion Criteria:

* Advanced/metastatic bladder cancer or advanced/metastatic cholangiocarcinoma.
* Prior receipt of a selective FGFR inhibitor.
* Current evidence of clinically significant corneal or retinal disorder.
* History of calcium and phosphate hemostasis disorder or systemic mineral imbalance with ectopic calcification of soft tissues.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2019-10-31 (Actual); Primary Completion 2020-06-12 (Actual); Study Completion 2020-06-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Incyte Medical Monitor, Study Director — Incyte Corporation
Locations (11):
- United States (11):
  - Compassionate Cancer Care Medical Group, Fountain Valley, California
  - Ocala Oncology Center, Ocala, Florida
  - Hawaii Cancer Care, Honolulu, Hawaii
  - Illinois Cancer Care, Peoria, Illinois
  - FMH James M Stockman Cancer Institute, Frederick, Maryland
  - New Jersey Cancer Care and Blood Disorders, Belleville, New Jersey
  - TriHealth, Cincinnati, Ohio
  - Sanford Cancer Center, Sioux Falls, South Dakota
  - Mary Crowley Cancer Center, Dallas, Texas
  - Oncology Consultants, Houston, Texas
  - Utah Cancer Specialists, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: Yes
Incyte shares data with qualified external researchers after a research proposal is submitted. These requests are reviewed and approved by a review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  The trial data availability is according to the criteria and process described on https://www.incyte.com/our-company/compliance-and-transparency
Supporting Information: Study Protocol, SAP
Time Frame: Data will be shared after the primary publication or 2 years after the study has ended for market authorized products and indications.
Access Criteria: Data from eligible studies will be shared with qualified researchers according to the criteria and process described in the Data Sharing section of the www.incyteclinicaltrials.com website. For approved requests, the researchers will be granted access to anonymized data under the terms of a data sharing agreement.
URL: https://www.incyte.com/our-company/compliance-and-transparency

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Approximately 50 participants were planned for enrollment. However, only 1 participant was enrolled in the study (assigned to Cohort A) and data was analyzed for safety. The study was closed for lack of enrollment in 2021.
Pre-assignment Details: A total of 1 participant (assigned to Cohort A) was enrolled in the study, received at least 1 dose of pemigatinib, and was included in the safety population. The participant withdrew consent after Cycle 2+. As a result, there was no efficacy evaluable population.
Groups:
- Cohort A: Participants With FGFR1-3 In-frame Fusions or FGFR2 Intron 17 Rearrangements; Cohort B: Participants With Known/Predicted Activating Point Mutations in FGFGR1-3: Participants will receive 13.5mg QD Pemigatinib
Period: Overall Study
Arm/Group | Cohort A: Participants With FGFR1-3 In-frame Fusions or FGFR2 Intron 17 Rearrangements | Cohort B: Participants With Known/Predicted Activating Point Mutations in FGFGR1-3
Started | 1 | 0
Completed | 0 | 0
Not Completed | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Population: No participants were enrolled in Cohort B.
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort A: Participants With FGFR1-3 In-frame Fusions or FGFR2 Intron 17 Rearrangements | Cohort B: Participants With Known/Predicted Activating Point Mutations in FGFGR1-3 | Total
Number analyzed (Participants) | 1 | 0 | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 1 | 0 | 1
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | NA — Due to low participant enrollment in this arm, data are not being reported, as doing so may risk participant identification. |  | NA — Total not calculated because data are not available (NA) in one or more arms.
  Male | NA — Due to low participant enrollment in this arm, data are not being reported, as doing so may risk participant identification. |  | NA — Total not calculated because data are not available (NA) in one or more arms.
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | NA — Due to low participant enrollment in this arm, data are not being reported, as doing so may risk participant identification. |  | NA — Total not calculated because data are not available (NA) in one or more arms.
  Asian | NA — Due to low participant enrollment in this arm, data are not being reported, as doing so may risk participant identification. |  | NA — Total not calculated because data are not available (NA) in one or more arms.
  Native Hawaiian or Other Pacific Islander | NA — Due to low participant enrollment in this arm, data are not being reported, as doing so may risk participant identification. |  | NA — Total not calculated because data are not available (NA) in one or more arms.
  Black or African American | NA — Due to low participant enrollment in this arm, data are not being reported, as doing so may risk participant identification. |  | NA — Total not calculated because data are not available (NA) in one or more arms.
  White | NA — Due to low participant enrollment in this arm, data are not being reported, as doing so may risk participant identification. |  | NA — Total not calculated because data are not available (NA) in one or more arms.
  More than one race | NA — Due to low participant enrollment in this arm, data are not being reported, as doing so may risk participant identification. |  | NA — Total not calculated because data are not available (NA) in one or more arms.
  Unknown or Not Reported | NA — Due to low participant enrollment in this arm, data are not being reported, as doing so may risk participant identification. |  | NA — Total not calculated because data are not available (NA) in one or more arms.

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate (ORR)
Description: Defined as the proportion of participants in each cohort who achieve a complete response (CR) or partial response (PR) based on Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST v1.1)
Time Frame: Up to approximately 6 months
Population: Due to low participant enrollment (n=1), efficacy analyses were not conducted.
Arm/Group | Cohort A: Participants With FGFR1-3 In-frame Fusions or FGFR2 Intron 17 Rearrangements | Cohort B: Participants With Known/Predicted Activating Point Mutations in FGFGR1-3
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Progression-free Survival (PFS)
Description: Defined as the time from first dose until progressive disease (per RECIST v1.1 or Response Assessment in Neuro-Oncology [RANO]) or death (whichever is first) in each cohort.
Time Frame: Up to approximately 6 months
Population: Due to low participant enrollment (n=1), efficacy analyses were not conducted.
Arm/Group | Cohort A: Participants With FGFR1-3 In-frame Fusions or FGFR2 Intron 17 Rearrangements | Cohort B: Participants With Known/Predicted Activating Point Mutations in FGFGR1-3
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Duration of Response (DOR)
Description: Defined as the time from the date of first assessment of CR or PR until the date of the first progressive disease (per RECIST v1.1 or RANO) or death (whichever is first) in each cohort.
Time Frame: Up to approximately 6 months
Population: Due to low participant enrollment (n=1), efficacy analyses were not conducted.
Arm/Group | Cohort A: Participants With FGFR1-3 In-frame Fusions or FGFR2 Intron 17 Rearrangements | Cohort B: Participants With Known/Predicted Activating Point Mutations in FGFGR1-3
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Disease Control Rate (DCR)
Description: Defined as the proportion of participants who achieved best overall response of CR, PR, or stable disease per RECIST v1.1 or RANO.
Time Frame: Up to approximately 6 months
Population: Due to low participant enrollment (n=1), efficacy analyses were not conducted.
Arm/Group | Cohort A: Participants With FGFR1-3 In-frame Fusions or FGFR2 Intron 17 Rearrangements | Cohort B: Participants With Known/Predicted Activating Point Mutations in FGFGR1-3
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Overall Survival (OS)
Description: Defined as the time from first dose of study drug to death of any cause in each cohort.
Time Frame: Up to approximately 6 months
Population: Due to low participant enrollment (n=1), efficacy analyses were not conducted.
Arm/Group | Cohort A: Participants With FGFR1-3 In-frame Fusions or FGFR2 Intron 17 Rearrangements | Cohort B: Participants With Known/Predicted Activating Point Mutations in FGFGR1-3
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Number of Treatment-related Adverse Events
Description: Adverse events reported for the first time or worsening of a pre-existing event after first dose of study drug/treatment.
Time Frame: Up to approximately 6 months
Population: Due to low participant enrollment (n=1), efficacy analyses were not conducted.
Arm/Group | Cohort A: Participants With FGFR1-3 In-frame Fusions or FGFR2 Intron 17 Rearrangements | Cohort B: Participants With Known/Predicted Activating Point Mutations in FGFGR1-3
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: May 2020 to June 2020
Description: Treatment-emergent adverse events, defined as adverse events that were either reported for the first time or the worsening of pre-existing events after the first dose of study drug until 30 days after the last dose of study drug, are reported for members of the Safety Population (all randomized participants who received at least one dose of study treatment).
Arm/Group | Cohort A: Participants With FGFR1-3 In-frame Fusions or FGFR2 Intron 17 Rearrangements | Cohort B: Participants With Known/Predicted Activating Point Mutations in FGFGR1-3
All-Cause Mortality (participants affected / at risk) | 0/1 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/1 | 0/0
Other Adverse Events (participants affected / at risk) | 1/1 | 0/0
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort A: Participants With FGFR1-3 In-frame Fusions or FGFR2 Intron 17 Rearrangements (N=1) | Cohort B: Participants With Known/Predicted Activating Point Mutations in FGFGR1-3 (N=0)
Blurred Vision (Eye disorders) | 1 (1) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Fatigue (General disorders) | 1 (1) | 0 (0)
Hyperphosphatemia (Metabolism and nutrition disorders) | 1 (2) | 0 (0)
Lower Back Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
The Sponsor made a decision unrelated to safety to halt study enrollment. Due to early termination of the study with only1 participant, no analysis of efficacy endpoints was done.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Following the first publication, the Institution and/or Principal Investigator may publish data or results from the Study, provided, however, that the Institution and/or Principal Investigator submits the proposed publication to the Sponsor for review at least sixty (60) days prior to the date of the proposed publication. Sponsor may remove from the proposed publication any information that is considered confidential and/or proprietary other than Study data and results.

DOCUMENTS (2):
  • Study Protocol (2019-06-14): https://cdn.clinicaltrials.gov/large-docs/23/NCT04003623/Prot_000.pdf
  • Statistical Analysis Plan (2021-06-21): https://cdn.clinicaltrials.gov/large-docs/23/NCT04003623/SAP_001.pdf